CLINICAL TRIAL: NCT00456092
Title: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Two Dose Regimens of CC-10004 in Subjects With Active Psoriatic Arthritis
Brief Title: Phase II Study of Apremilast (CC-10004) in Adults With in Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-001
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; ACR; PASI; DAS; pharmacokinetic; biopsy
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apremilast 40 mg QD (Experimental): Participants received 40 mg apremilast orally once a day (QD) for 12 weeks in the Treatment Phase. Participants who entered the Extension Phase continued to receive 40 mg apremilast QD for an additional 12 weeks.
  The dose of apremilast was titrated starting at 10 mg QD during Days 1 to 3 followed by 20 mg QD during Days 4 to 7 and then 40 mg QD thereafter. A single dose reduction to 20 mg per day was allowed for participants who experienced intolerable adverse effects from study medication.
  Interventions: Drug: Apremilast
- Apremilast 20 mg BID (Experimental): Participants received 20 mg apremilast orally twice a day (BID) for 12 weeks in the Treatment Phase. Participants who entered the Extension Phase continued to receive 20 mg apremilast BID for an additional 12 weeks. The dose of apremilast was titrated starting at 10 mg QD during Days 1 to 3 followed by 20 mg QD during Days 4 to 7 and then 20 mg BID thereafter. A single dose reduction to 20 mg per day was allowed for participants who experienced intolerable adverse effects from study medication.
  Interventions: Drug: Apremilast
- Placebo (Placebo Comparator): Participants received matching placebo to apremilast orally BID for 12 weeks during the Treatment Phase. Participants who entered the Extension Phase were re-randomized on Day 85 to receive either 40 mg apremilast QD or 20 mg apremilast BID for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Capsules for oral administration
  Other Names: CC-10004; Otezla®
  Arms: Apremilast 20 mg BID; Apremilast 40 mg QD
Drug: Placebo — Capsules for oral administration
  Arms: Placebo

SUMMARY:
This study is to look at the preliminary efficacy and safety of 2 dose regimens of apremilast (20 mg twice a day and 40 mg once a day) versus placebo in patients with active psoriatic arthritis.

DETAILED DESCRIPTION:
Prior to the implementation of Amendment 1/UK3 the study consisted of 3 phases - pre-randomization up to 35 days, up to 84 days placebo-controlled treatment and a 28-day observational follow up. After the implementation of Amendment 1/UK3, the study consisted of 4 phases - pre-randomization up to 35 days, up to 84 days treatment in the placebo controlled treatment phase, up to 84 days treatment in the active treatment extension phase and a 28 day follow up. Participants who completed the treatment phase prior to implementation of amendment 1/UK3 did not have the option of entering the extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psoriatic arthritis (Moll and Wright Criteria), including symmetrical or asymmetrical peripheral joint involvement for at least 6 months
* Active psoriatic arthritis at the time of screening and baseline as defined by: 3 or more swollen joints AND 3 or more tender joints
* Negative rheumatoid factor (RF)
* If using methotrexate, be on methotrexate for at least 168 days (24 weeks) and be on a stable dose for at least 56 days prior to screening and throughout the study
* If using oral corticosteroids, be on a stable dose of prednisone ≤ 10 mg/day or equivalent for at least 28 days prior to screening and throughout the study
* If using nonsteroidal anti-inflammatory drug (NSAID) therapy, be on a stable dose for at least 14 days prior to screening and throughout the study
* Must meet the following laboratory criteria:

  * Hemoglobin ≥ 9 g/dL
  * Hematocrit ≥ 27%
  * White blood cell (WBC) count ≥ 3000/μL (≥ 3.0 X 10^9/L) and < 20,000/μL (< 20 X 10^9/L)
  * Neutrophils ≥ 1500 /μL (≥ 1.5 X 10^9/L)
  * Platelets ≥ 100,000 /μL (≥ 100 X 10^9/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * Total bilirubin ≤ 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) ≤ 1.5x upper limit of normal (ULN)
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO adequate forms of contraception while on study medication. A FCBP must agree to have pregnancy tests every 28 days while on study medication
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP while on study medication and for at least 84 days after taking the last dose of study medication

Exclusion Criteria:

History of any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases

* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or lactating female
* History of active Mycobacterium tuberculosis infection (any subspecies) within 3 years prior to the screening visit. Infections that occurred > 3 years prior to entry must have been effectively treated.
* History of incompletely treated latent Mycobacterium tuberculosis infection (as indicated by a positive Purified Protein Derivative [PPD] skin test or in vitro test [T SPOT®.TB, QuantiFERON Gold®])
* Clinically significant abnormality on the chest x-ray (CXR) at screening
* Current erythrodermic, guttate, or pustular forms of psoriasis
* History of infected joint prosthesis within the past 5 years
* Systemic therapy for psoriasis and/or psoriatic arthritis (except for methotrexate, ≤ 10 mg/day prednisone or equivalent, and NSAIDs) including, but not limited to, sulfasalazine, leflunomide, chloroquine, hydroxychloroquine, gold compounds, parenteral corticosteroids (including intra-articular), penicillamine, cyclosporine, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, tacrolimus, azathioprine, and fumaric acid esters within 28 days of randomization and throughout the study
* Topical therapy for the treatment of psoriasis including, but not limited to topical steroids, topical vitamin A or D analog preparations, tacrolimus, pimecrolimus, or anthralin within 14 days of randomization (Note: Topical background therapy for treatment of psoriasis is allowed, except within 24 hours of a study visit, as follows: mild or moderate potency corticosteroids for treatment of the palms, face, scalp, axillae, plantar surfaces, and groin in accordance with the manufacturer's suggested usage. Nonmedicated emollients [eg, Eucerin®] and tar shampoo are also allowed.)
* Phototherapy (ultraviolet light A [UVA], narrow-band ultraviolet light B [NB-UVB], psoralens and long-wave ultraviolet radiation [PUVA]) within 28 days prior to randomization
* Etanercept use within 56 days prior to randomization
* Adalimumab, efalizumab, or infliximab use within 84 days prior to randomization
* Alefacept use within 168 days (24 weeks) prior to randomization
* Use of intra-articular corticosteroids within 28 days prior to randomization
* Use of any investigational medication within 28 days prior to randomization or 5 half-lives if known (whichever is longer)
* Any clinically significant abnormality on 12-lead electrocardiogram (ECG) at screening
* High-risk factor(s) for, or a history of, human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus infection
* History of malignancy within previous 5 years (except for treated basal-cell skin carcinoma(s) and/or fewer than 3 treated squamous-cell skin carcinomas)
* Evidence of skin conditions at the time of screening visit that would interfere with evaluations of the effect of study medication on psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2007-03-05 (Actual); Primary Completion 2009-05-09 (Actual); Study Completion 2009-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- Belgium (4):
  - CHU Brugmann, Brussels
  - Universiteit Hasselt, Diepenbeek
  - University Hospital, Leuven
  - Jan Palfijn Ziekenhuis, Merksem
- Canada (15):
  - The Arthritis Research Centre of Canada, Vancouver, British Columbia
  - Victoria, British Columbia
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Burlington Rheumatology and Osteoporosis Clinic, Burlington, Ontario
  - MAC Research Inc., Hamilton, Ontario
  - K-W Musculoskeletal Research Inc., Kitchener, Ontario
  - Credit Valley Rheumatology, Mississauga, Ontario
  - Arthritis Program Research Group Inc, Newmarket, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Center for Prognosis Studies in the Rheumatic Diseases University Health Network, Toronto Western Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Probity Medical, Waterloo, Ontario
  - Clinical Research and Arthritis Centre, Windsor, Ontario
  - West Island Rheumatology Research Associates, Pointe-Claire, Quebec
  - Saskatoon Osteoporosis Center, Saskatoon, Saskatchewan
- Germany (12):
  - Capio Franz von Prümmer Klinik, Bad Brückenau
  - Free University of Berlin, Berlin
  - Universitaetsklinik Koeln, Cologne
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Klinikum Eilbek, Hamburg
  - Universitaet Heidelberg, Heidelberg
  - Rheumazentrum Ruhrgebiet, Herne
  - Universitaet Leipzig, Leipzig
  - Universitaetsklinikum Leipzig, Leipzig
  - University of Munich, Munich
  - Klinikum der Universität Munster, Münster
  - Friedrich-Alexander University, Erlangen, Nuremberg
- Netherlands (3):
  - Leiden University Medical Centre, Leiden
  - Radboud University, Nijmegen
  - Hagaziekenhuis, The Hague
- United Kingdom (4):
  - Hope Hospital, Salford, Manchester
  - Haywood Hospital, Stoke-on-Trent, Staffs
  - Chapel Allerton Hospital, Leeds
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Schett G, Wollenhaupt J, Papp K, Joos R, Rodrigues JF, Vessey AR, Hu C, Stevens R, de Vlam KL. Oral apremilast in the treatment of active psoriatic arthritis: results of a multicenter, randomized, double-blind, placebo-controlled study. Arthritis Rheum. 2012 Oct;64(10):3156-67. doi: 10.1002/art.34627. PMID 22806399
- [Result] Strand V, Schett G, Hu C, Stevens RM. Patient-reported Health-related Quality of Life with apremilast for psoriatic arthritis: a phase II, randomized, controlled study. J Rheumatol. 2013 Jul;40(7):1158-65. doi: 10.3899/jrheum.121200. Epub 2013 Apr 15. PMID 23588944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 38 sites in Canada, Belgium, Germany, the Netherlands, and the United Kingdom.
Pre-assignment Details: Participants were randomized 1:1:1 to either apremilast 40 mg once daily, 20 mg twice daily, or placebo. On Day 85 participants originally randomized to placebo were re-randomized to receive apremilast; participants randomized to apremilast continued on the same dose regimen. Randomization was stratified based on methotrexate use at baseline.
Groups:
- Placebo/Apremilast 40 mg QD: Participants who received placebo during the Treatment Phase then received 40 mg apremilast orally QD for 12 weeks during the Extension Phase. The dose of apremilast was titrated starting at 10 mg QD during Days 85 to 87 followed by 20 mg QD during Days 88 to 91 and then 40 mg QD thereafter. A single dose reduction to 20 mg per day was allowed for participants who experienced intolerable adverse effects from study medication.
- Placebo/Apremilast 20 mg BID: Participants who received placebo during the Treatment Phase then received 20 mg apremilast orally BID for 12 weeks during the Extension Phase. The dose of apremilast was titrated starting at 10 mg QD during Days 85 to 87 followed by 20 mg QD during Days 88 to 91 and then 20 mg BID thereafter. A single dose reduction to 20 mg per day was allowed for participants who experienced intolerable adverse effects from study medication.
Period: Extension Phase
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Started | 46 (The Extension Phase was only open to participants enrolled after amendment 1 was in effect.) | 40 (The Extension Phase was only open to participants enrolled after amendment 1 was in effect.) | 0 | 20 (The Extension Phase was only open to participants enrolled after amendment 1 was in effect.) | 20 (The Extension Phase was only open to participants enrolled after amendment 1 was in effect.)
Completed | 35 | 36 | 0 | 19 | 13
Not Completed | 11 | 4 | 0 | 1 | 7
Not completed — Grade 2 or Greater AE | 2 | 2 | 0 | 0 | 2
Not completed — Flare of Psoriatic Arthritis | 1 | 0 | 0 | 0 | 1
Not completed — Worsening / Not Responding to Study Drug | 3 | 1 | 0 | 0 | 2
Not completed — Withdrew Consent | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1
Not completed — Other | 2 | 0 | 0 | 1 | 1
Period: Treatment Phase (12 Weeks)
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Started | 67 | 69 | 68 | 0 | 0
Completed | 60 | 55 | 50 | 0 | 0
Not Completed | 7 | 14 | 18 | 0 | 0
Not completed — Grade 2 or Greater Adverse Event (AE) | 3 | 4 | 2 | 0 | 0
Not completed — AEs not Included in NCI Terminology | 1 | 2 | 0 | 0 | 0
Not completed — Intolerability of the Study Drug | 2 | 0 | 0 | 0 | 0
Not completed — Flare of Psoriasis | 0 | 1 | 2 | 0 | 0
Not completed — Flare of Psoriatic Arthritis | 0 | 3 | 3 | 0 | 0
Not completed — Worsening / Not Responding to Study Drug | 0 | 2 | 7 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Apremilast 40 mg QD: Participants received 40 mg apremilast once daily (QD) for 12 weeks in the Treatment Phase.
- Apremilast 20 mg BID: Participants received 20 mg apremilast twice a day (BID) for 12 weeks in the Treatment Phase.
- Placebo: Participants received matching placebo to apremilast for 12 weeks during the Treatment Phase.
- Total: Total of all reporting groups
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo | Total
Number analyzed (Participants) | 67 | 69 | 68 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.17) | 50.9 (12.58) | 51.1 (10.80) | 50.6 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 36 | 97
  Male | 32 | 43 | 32 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 62 | 67 | 68 | 197
  Black | 1 | 0 | 0 | 1
  Hispanic | 1 | 0 | 0 | 1
  Asian/Pacific Islander | 2 | 1 | 0 | 3
  American Indian/Alaska Native | 0 | 0 | 0 | 0
  Other | 1 | 1 | 0 | 2
Psoriatic Arthritis Disease Category [Count of Participants; unit: Participants]
  Asymmetrical Oligoarthritis | 26 | 21 | 20 | 67
  Predominant Spondylitis | 4 | 3 | 2 | 9
  Symmetric Polyarthritis | 32 | 36 | 39 | 107
  Arthritis Mutilans | 2 | 0 | 5 | 7
  Predominant Distal Interphalgeal Involvement | 2 | 9 | 2 | 13
  Missing/Unknown | 1 | 0 | 0 | 1
Duration of Psoriatic Arthritis [Mean (Standard Deviation); unit: years] | 7.6 (8.73) | 8.4 (9.77) | 7.3 (6.74) | 7.8 (8.48)
Pain/Tender Joint Score [Mean (Standard Deviation); unit: joints] — The number of tender joints (joints with scores of 1 to 3), rated on a scale of 0 (no pain/tenderness) to 3 (severe pain - tender, winced, withdrew). The joint count included the 68 joints routinely utilized in the American College of Rheumatology (ACR) joint count for evaluation of rheumatoid arthritis, plus 10 additional joints often involved in psoriatic arthritis (the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers) for a total of 78 joints.
  joints | 23.2 (17.63) | 20.6 (15.90) | 21.3 (15.55) | 21.7 (16.33)
Swollen Joint Score [Mean (Standard Deviation); unit: joints] — The number of swollen joints noted by the examiner. The joint count included the 66 joints routinely utilized in the American College of Rheumatology (ACR) joint count for evaluation of rheumatoid arthritis, plus 10 additional joints often involved in psoriatic arthritis (the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers) for a total of 76 joints.
  joints | 8.4 (4.94) | 10.6 (9.88) | 9.5 (9.68) | 9.5 (8.51)
Psoriasis Severity [Count of Participants; unit: Participants] — Psoriasis severity was assessed by the Investigator.
  Participants
    None | 2 | 7 | 12 | 21
    Mild | 41 | 47 | 40 | 128
    Moderate | 20 | 15 | 11 | 46
    Severe | 4 | 0 | 5 | 9
Duration of Psoriasis [Mean (Standard Deviation); unit: years] | 18.3 (13.62) | 15.5 (11.66) | 15.8 (13.22) | 16.5 (12.85)
Methotrexate Use [Count of Participants; unit: Participants]
  Yes | 30 | 30 | 29 | 89
  No | 37 | 39 | 39 | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Modified American College of Rheumatology 20% (ACR 20) Response at Week 12
Description: A modified American College of Rheumatology 20% (ACR 20) response was defined as a participant who met the following 3 criteria for improvement from Baseline: • ≥ 20% improvement in 78 tender joint count (includes 10 additional joints often involved in psoriatic arthritis: the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers); • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. Participants with no post-baseline ACR scores were considered non-responders.
Time Frame: Baseline and Week 12
Population: The intent-to-treat (ITT) population which consisted of all randomized participants with at least one of the ACR components assessed at baseline. Last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 40 mg QD: Participants received 40 mg apremilast once daily (QD) for 12 weeks during the Treatment Phase.
- Apremilast 20 mg BID: Participants received 20 mg apremilast twice a day (BID) for 12 weeks during the Treatment Phase.
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 35.8 | 43.5 | 11.8
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.002, Chi-squared, Corrected — A p-value < 0.025 (2-sided) is considered statistically significant, after adjusting for two treatment comparisons using the Bonferroni procedure; Odds Ratio (OR) = 4.190, 95% CI 2-sided [1.72 to 10.20]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p < 0.001, Chi-squared, Corrected — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.770, 95% CI 2-sided [2.40 to 13.88]

2. Secondary Outcome: Number of Participants With Adverse Events During the Treatment Phase
Description: The severity of each adverse event (AE) was graded based upon the participant's symptoms according to National Cancer Institute (NCI) Common Toxicity Criteria (CTCAE, Version 3.0), on a scale from 1 (Mild AE) to 5 (Death due to AE). Severe AEs are defined as NCI CTCAE grade 3 or higher. AEs related to study drug are those determined by the investigator as suspected to be related to study drug where a temporal relationship of the adverse event to study drug administration made a causal relationship possible, and other medications, therapeutic interventions, or underlying conditions did not provide a sufficient explanation for the observed event. A serious adverse event (SAE) is any AE which: - Resulted in death - Was life-threatening - Required inpatient hospitalization or prolongation of existing hospitalization - Resulted in persistent or significant disability/incapacity - Was a congenital anomaly/birth defect - Constituted an important medical event.
Time Frame: 12 weeks
Population: The safety population which consisted of all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
Participants
  All adverse events | 58 | 59 | 55
  Adverse events related to study drug | 27 | 26 | 26
  Severe adverse events | 5 | 4 | 6
  Severe adverse events related to study drug | 1 | 1 | 1
  Serious adverse events | 0 | 4 | 4
  Serious adverse events related to study drug | 0 | 0 | 1
  Discontinued study drug due to adverse event | 6 | 10 | 7
  Discontinued due to AE related to study drug | 5 | 4 | 1

3. Secondary Outcome: Percentage of Participants With a Psoriatic Arthritis Response Criteria (PsARC) Response at Week 12
Description: A PsARC response is defined as improvement from Baseline in at least 2 of the following 4 measures, at least 1 of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures, according to the following: • At least 30% improvement in the 78 tender joint count, • At least 30% improvement in the 76 swollen joint count, • At least 20% improvement in the patient global assessment of disease activity, measured on a 100 mm visual analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • At least 20% improvement in the physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Participants with no post-baseline PsARC scores were considered non-responders.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 50.7 | 52.2 | 22.1

4. Secondary Outcome: Percentage of Participants With a Modified ACR 50 Response at Week 12
Description: A modified American College of Rheumatology 50% (ACR 50) response was defined as a participant who met the following 3 criteria for improvement from Baseline: • ≥ 50% improvement in 78 tender joint count (includes 10 additional joints often involved in psoriatic arthritis: the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers); • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. Participants with no post-baseline ACR scores were considered non-responders.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 13.4 | 17.4 | 2.9
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.056, Chi-squared, Corrected; Odds Ratio (OR) = 5.120, 95% CI 2-sided [1.06 to 24.67]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.012, Chi-squared, Corrected; Odds Ratio (OR) = 6.950, 95% CI 2-sided [1.49 to 32.35]

5. Secondary Outcome: Percentage of Participants With a Modified ACR 70 Response at Week 12
Description: A modified American College of Rheumatology 70% (ACR 70) response was defined as a participant who met the following 3 criteria for improvement from Baseline: • ≥ 70% improvement in 78 tender joint count (includes 10 additional joints often involved in psoriatic arthritis: the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers); • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-reactive protein. Participants with no post-baseline ACR scores were considered non-responders.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 7.5 | 5.8 | 1.5
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.204, Chi-squared, Corrected; Odds Ratio (OR) = 5.400, 95% CI 2-sided [0.61 to 47.54]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.371, Chi-squared, Corrected; Odds Ratio (OR) = 4.120, 95% CI 2-sided [0.45 to 37.88]

6. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response Based on Disease Activity Score (DAS28)-CRP(4) at Week 12
Description: The DAS28 measures the severity of disease at a specific time. DAS28-CRP(4) is derived from the following 4 variables: • 28 tender joint count, (TJC; does not include the DIP joints, the hip joint, or the joints below the knee) • 28 swollen joint count (SJC) • C-reactive protein (CRP) • Patient's global assessment of disease activity (GH) according to the formula: DAS28-CRP(4) = 0.56*√(TJC28) + 0.28*(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96. DAS28 scores range from 0 to 9.4, where higher scores indicate more disease activity. A EULAR response reflects an improvement in disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 > 1.2 from Baseline and a DAS28 score ≤ 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 > 0.6 and ≤ 1.2 and a DAS28 score ≤ to 5.1 or, • an improvement (decrease) in the DAS28 > 1.2 and a DAS28 score > 3.2
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; LOCF imputation was used. Participants with no baseline or post-baseline DAS28-CRP(4) scores were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 49.3 | 55.1 | 38.2
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.264, Chi-squared, Corrected; Odds Ratio (OR) = 1.568, 95% CI 2-sided [0.79 to 3.11]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.071, Chi-squared, Corrected; Odds Ratio (OR) = 1.980, 95% CI 2-sided [1.00 to 3.91]

7. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response Based on DAS28-CRP(3) at Week 12
Description: The DAS28 measures the severity of disease at a specific time. DAS28-CRP(3) is derived from the following 3 variables: • 28 tender joint count, (does not include the DIP joints, the hip joint, or the joints below the knee) • 28 swollen joint count • C-reactive protein (CRP) according to the formula: DAS28-CRP(3) = [0.56*√(TJC28) + 0.28*√(SJC28) + 0.36*ln(CRP+1)] * 1.10 + 1.15. DAS28 scores range from 0 to 9.4, where higher scores indicate more disease activity. A EULAR response reflects an improvement in disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 > 1.2 from Baseline and attainment of a DAS28 score ≤ 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 > 0.6 and ≤ 1.2 and a DAS28 score ≤ to 5.1 or, • an improvement (decrease) in the DAS28 > 1.2 and a DAS28 score > 3.2
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; LOCF imputation was used. Participants with no baseline or post-baseline DAS28-CRP(3) scores were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 50.7 | 44.9 | 44.1
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.549, Chi-squared, Corrected; Odds Ratio (OR) = 1.305, 95% CI 2-sided [0.66 to 2.57]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; Odds Ratio (OR) = 1.033, 95% CI 2-sided [0.53 to 2.03]

8. Secondary Outcome: Percentage of Participants With DAS28-CRP(4) Score of Mild Disease Activity or In Remission at Week 12
Description: The DAS28-CRP(4) measures the severity of disease derived from the following 4 variables: • 28 tender joint count, (does not include the DIP joints, the hip joint, or the joints below the knee) • 28 swollen joint count • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28-CRP(4) scores range from 0 to 9.4, where higher scores indicate more disease activity. Mild disease severity is defined as a DAS28-CRP(4) score of ≤ 3.2. In remission is defined as a DAS28-CRP(4) score of ≤ 2.6.
Time Frame: Week 12
Population: Intent-to-treat population; LOCF imputation was used. Participants with no post-baseline DAS28-CRP(4) scores were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 38.8 | 33.3 | 23.5
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.083, Chi-squared, Corrected; Odds Ratio (OR) = 2.060, 95% CI 2-sided [0.98 to 4.34]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.279, Chi-squared, Corrected; Odds Ratio (OR) = 1.630, 95% CI 2-sided [0.77 to 3.44]

9. Secondary Outcome: Percentage of Participants With DAS28-CRP(3) Score of Mild Disease Activity or In Remission at Week 12
Description: The DAS28-CRP(3) measures the severity of disease derived from the following 3 variables: • 28 tender joint count (does not include the DIP joints, the hip joint, or the joints below the knee) • 28 swollen joint count • C-reactive protein (CRP) DAS28-CRP(3) scores range from 0 to 9.4, where higher scores indicate more disease activity. Mild disease severity is defined as a DAS28-CRP(3) score of ≤ 3.2. In remission is defined as a DAS28-CRP(3) score of ≤ 2.6.
Time Frame: Week 12
Population: Intent-to-treat population; LOCF imputation was used. Participants with no post-baseline DAS28-CRP(3) scores were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants | 40.3 | 34.8 | 33.8
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.548, Chi-squared, Corrected; Odds Ratio (OR) = 1.320, 95% CI 2-sided [0.66 to 2.66]
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; Odds Ratio (OR) = 1.040, 95% CI 2-sided [0.52 to 2.11]

10. Secondary Outcome: Number of Participants Who Withdrew Prematurely Due to Lack of Efficacy
Description: The number of participants who withdrew prematurely from the treatment phase due to lack of efficacy, including flare of psoriasis, flare of psoriatic arthritis or worsening or not responding to study treatment.
Time Frame: Baseline to Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
Participants | 0 | 6 | 12

11. Secondary Outcome: Number of Participants With Adverse Events Leading to a Dose Reduction
Description: The number of participants who were dose reduced during the treatment phase due to adverse events.
Time Frame: Baseline to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
Participants | 4 | 4 | 0

12. Secondary Outcome: Maximal ACR Response During the Treatment Phase
Description: The ACR-N index score was calculated for each participant at each time point in the study according to the following definition: ACR-N = the lowest of the following 3 values: - percent improvement from Baseline in the 76 swollen joint count, - percent improvement from Baseline in the 78 tender joint count - median percent improvement from Baseline in the following 5 measures ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. The maximal ACR-N for each participant during the 12-week treatment period was calculated, and represents the maximal ACR response achieved.
Time Frame: ACR was measured at Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: Intent-to-treat population with non-missing ACR data
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 65 | 67 | 65
percent improvement | 22.3 (56.45) | 24.2 (37.63) | 10.7 (35.42)
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.136, ANOVA; ANOVA model with treatment as the factor; Treatment Difference = 11.58 — Treatment Difference = Apremilast 20 mg BID - Placebo
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.080, ANOVA; ANOVA model with treatment as the factor; Treatment Difference = 13.53 — Treatment Difference = Apremilast 20 mg BID - Placebo

13. Secondary Outcome: Time to ACR 20 Response During the Treatment Phase
Description: The Kaplan-Meier estimates of time to ACR 20 response was calculated for participants who had an ACR 20 response at any time during the treatment phase.
Time Frame: Baseline to Week 12
Population: Intent-to-treat population with an ACR 20 response during the treatment phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 37 | 43 | 31
days | 29.0 [29.0 to 43.0] | 30.0 [29.0 to 57.0] | 29.0 [20.0 to 47.0]
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.650, Chi-squared; Hazard Ratio (HR) = 0.950, 95% CI 2-sided [0.745 to 1.211] — Based on a proportional hazards model comparing the hazard functions associated with the treatment and placebo
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.283, Chi-squared; Hazard Ratio (HR) = 1.265, 95% CI 2-sided [0.791 to 2.024] — Based on a proportional hazards model comparing the hazard functions associated with the treatment and placebo

14. Secondary Outcome: Time to ACR 50 Response During the Treatment Phase
Description: The Kaplan-Meier estimates of time to ACR 50 response was calculated for participants who had an ACR 50 response at any time during the treatment phase.
Time Frame: Baseline to Week 12
Population: Intent-to-treat population who had an ACR 50 response during the treatment phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 17 | 18 | 5
days | 43.0 [29.0 to 61.0] | 57.5 [56.0 to 72.0] | 15.0 [14.0 to 73.0]
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.253, Chi-squared; Hazard Ratio (HR) = 1.337, 95% CI 2-sided [0.791 to 2.260] — Based on a proportional hazards model comparing the hazard functions associated with the treatment and placebo
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.026, Chi-squared; Hazard Ratio (HR) = 3.023, 95% CI 2-sided [1.059 to 8.630] — Based on a proportional hazards model comparing the hazard functions associated with the treatment and placebo

15. Secondary Outcome: Time to ACR 70 Response During the Treatment Phase
Description: The Kaplan-Meier estimates of time to ACR 70 response was calculated for participants who had an ACR 70 response at any time during the treatment phase.
Time Frame: Baseline to Week 12
Population: Intent-to-treat population with an ACR 70 response during the treatment phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 7 | 5 | 2
days | 62.0 [47.0 to 85.0] | 57.0 [43.0 to 85.0] | 58.0 [31.0 to 85.0]
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.984, Chi-squared; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.457 to 2.215] — Based on a proportional hazards model comparing the hazard functions associated with the treatment and placebo
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.836, Chi-squared; Hazard Ratio (HR) = 0.872, 95% CI 2-sided [0.158 to 4.797] — Based on a proportional hazards model comparing the hazard functions associated with the treatment and placebo

16. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 12
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated on a scale from 0 (no dactylitis) to 3 (severe dactylitis). The dactylitis severity score is the sum of the individual scores for each digit and ranges from 0 to 60.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; participants with a baseline value and at least 1 post-baseline value in the treatment period are included; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 67 | 67
units on a scale | -0.9 (2.39) | -1.2 (3.11) | -0.2 (3.75)

17. Secondary Outcome: Percentage of Participants With Enthesitis
Description: Enthesitis is inflammation of the entheses, the sites where tendons or ligaments insert into the bone. Enthesitis is characterized by swelling, pain, and tenderness around the calcaneous, and occasionally by effusion in the bursa associated with this joint. The enthesitis assessment is an evaluation of inflammation at the insertions of the Achilles tendon into the calcaneous and of the plantar fascia into the calcaneous. Inflammation at 1 or more insertions on either the right or left side constituted a positive assessment.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 68
percentage of participants
  Achilles tendon into the calcaneous: Baseline | 22.4 | 21.7 | 35.3
  Achilles tendon into the calcaneous: Week 12 | 20.9 | 17.4 | 17.6
  Plantar fascia into the calcaneous: Baseline | 26.9 | 26.1 | 14.7
  Plantar fascia into the calcaneous: Week 12 | 19.4 | 21.7 | 17.6

18. Secondary Outcome: Time to Relapse of Psoriatic Arthritis During the Observational Follow-up Phase
Description: Relapse of psoriatic arthritis was defined as a 50% loss of the maximal ACR improvement during the Observation Phase in participants who received apremilast and achieved at least an ACR 20 at their Final Treatment Phase/Early Termination Visit. The time to relapse during the Observational Phase was calculated from the time of maximum ACR reduction and from the date of the Final Treatment Phase visit. Participants classified as responders who did not relapse were censored at the day of the last follow-up.
Time Frame: From Week 12 to end of 28-day observational follow-up (1) and from the date of maximal ACR during the 12-week Treatment Phase until the end of the 28-day observational follow-up phase (2).
Population: Participants who received apremilast and with an ACR 20 response at the Week 12 (or Early Termination) visit who did not enroll in the Extension Phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID
Number analyzed (Participants) | 7 | 11
days
  1. From Week 12 | 16.0 [15.0 to 29.0] | 15.0 [14.0 to 29.0]
  2. From Date of Maximal ACR Response | 43.0 [34.0 to 73.0] | 29.0 [22.0 to 43.0]

19. Secondary Outcome: Number of Participants Who Relapsed During the Observational Follow-up Phase
Description: Relapse of psoriatic arthritis was defined as a 50% loss of the maximal ACR improvement during the Observation Phase in participants who received apremilast and achieved at least an ACR 20 at their Final Treatment Phase/Early Termination Visit.
Time Frame: 28-day observational follow-up period following Week 12
Population: Participants who received apremilast with an ACR 20 response at the Week 12 (or Early Termination) visit who did not enroll in the Extension Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID
Number analyzed (Participants) | 7 | 11
Participants | 5 | 9

20. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Summary Physical and Mental Component Scores at Week 12
Description: The Medical Outcome SF 36-Item Health Survey, Version 2 is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The summary physical health score included the following subscales: physical functioning, role-physical, bodily pain, and general health. The summary mental health score included other subscales: vitality, social functioning, role-emotional, and mental health. Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10, where higher scores are associated with better functioning/quality of life. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale. A higher change from baseline indicates an improvement in better health results or functioning.
Time Frame: Baseline and Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 65 | 64 | 61
units on a scale
  Mental Component | 1.0 (8.01) | 3.4 (7.18) | -0.8 (8.39)
  Physical Component | 2.1 (5.94) | 2.4 (7.89) | 0.8 (6.24)
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Mental Component; Test type: Superiority; p = 0.308, ANOVA; ANOVA model including treatment group, methotrexate use, and baseline score; Adjusted Mean Difference = 1.4 — Adjusted mean difference (Apremilast-Placebo) was based on the ANOVA model described above
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Mental Component; Test type: Superiority; p = 0.003, ANOVA; ANOVA model including treatment group, methotrexate use, and baseline score; Adjusted Mean Difference = 4.1 — Adjusted mean difference (Apremilast-Placebo) was based on the ANOVA model described above
Statistical Analysis 3: Comparison: Apremilast 40 mg QD vs Placebo; Physical Component; Test type: Superiority; p = 0.182, ANOVA; ANOVA model including treatment group, methotrexate use, and baseline score; Adjusted Mean Difference = 1.6 — Adjusted mean difference (Apremilast-Placebo) was based on the ANOVA model described above
Statistical Analysis 4: Comparison: Apremilast 20 mg BID vs Placebo; Physical Component; Test type: Superiority; p = 0.026, ANOVA; ANOVA model including treatment group, methotrexate use, and baseline score; Adjusted Mean Difference = 2.7 — Adjusted mean difference (Apremilast-Placebo) was based on the ANOVA model described above

21. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 12
Description: The DLQI is a validated, self-administered, 10-item questionnaire that measures the impact of skin disease on participants' quality of life, based on recall over the past week. Domains include symptoms, feelings, daily activities, leisure, work, personal relationships, and treatment. Each question is answered on a scale from 0 (not at all) to 3 (very much). The total score ranges from 0 to 30 where a higher score indicates that a participant's dermatological condition has a greater impact on their daily life.
Time Frame: Baseline and Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 67 | 64
units on a scale | -2.6 (5.96) | -1.8 (4.29) | -0.3 (4.82)
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.016, ANOVA; ANOVA model using treatment group, methotrexate use, and interaction of treatment group and methotrexate use as factors; Adjusted Mean Difference = -2.1 — The adjusted mean difference (Apremilast-Placebo) is based on an ANOVA model described above
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.105, ANOVA; ANOVA model using treatment group, methotrexate use, and interaction of treatment group and methotrexate use as factors; Adjusted Mean Difference = -1.4 — The adjusted mean difference (Apremilast-Placebo) is based on an ANOVA model described above

22. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The HAQ-DI is a self-administered instrument consisting of 20 questions in eight categories of functioning which represent a comprehensive set of functional activities - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item asks over the past week whether a particular task can be performed. For each item, there is a four-level difficulty scale that is scored from 0 to 3, representing normal (no difficulty) (0), some difficulty (1), much difficulty (2), and unable to do (3). The eight category scores are averaged into an overall HAQ-DI score on a scale from zero (no disability) to three (completely disabled).
Time Frame: Baseline and Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 67
units on a scale | -0.2 (0.39) | -0.2 (0.35) | -0.1 (0.39)

23. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy for Fatigue (FACIT-F) at Week 12
Description: The FACIT-Fatigue is a 13 item self-administered questionnaire that assesses both the physical and functional consequences of fatigue based on recall during the past 7 days. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The total score ranges from 0 to 52 with higher scores representing less fatigue.
Time Frame: Baseline and Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo
Number analyzed (Participants) | 67 | 67 | 64
units on a scale | 4.3 (9.46) | 4.1 (8.78) | 0.5 (8.03)
Statistical Analysis 1: Comparison: Apremilast 40 mg QD vs Placebo; Test type: Superiority; p = 0.028, ANOVA; ANOVA model with treatment, methotrexate use, and interaction of treatment group and methotrexate use as factors and baseline score as the covariate; Adjusted Mean Difference = 3.3 — The adjusted mean difference (Apremilast-Placebo) is based on an ANOVA model described above
Statistical Analysis 2: Comparison: Apremilast 20 mg BID vs Placebo; Test type: Superiority; p = 0.004, ANOVA; ANOVA model with treatment, methotrexate use, and interaction of treatment group and methotrexate use as factors with baseline score as the covariate; Adjusted Mean Difference = 4.3 — The adjusted mean difference (Apremilast-Placebo) is based on an ANOVA model described above

24. Secondary Outcome: Number of Participants With Adverse Events During the Extension Phase
Description: as for outcome 2
Time Frame: Weeks 12 to 24 (Extension Phase)
Population: The safety population; participants who entered the Extension Phase.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast 40 mg QD: Participants who received apremilast 40 mg QD during the Treatment Phase continued to receive apremilast 40 mg QD for an additional 12 weeks during the Extension Phase.
- Apremilast 20 mg BID: Participants who received apremilast 20 mg BID during the Treatment Phase continued to receive apremilast 20 mg BID for an additional 12 weeks during the Extension Phase.
- Placebo/Apremilast 40 mg QD: Participants who received placebo during the Treatment Phase then received 40 mg apremilast orally QD for 12 weeks during the Extension Phase.
- Placebo/Apremilast 20 mg BID: Participants who received placebo during the Treatment Phase then received 20 mg apremilast orally BID for 12 weeks during the Extension Phase.
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
Participants
  All adverse events | 30 | 29 | 16 | 11
  Adverse events related to study drug | 12 | 8 | 4 | 4
  Severe adverse events | 5 | 3 | 3 | 4
  Serious adverse events | 2 | 3 | 1 | 1
  Serious adverse events related to study drug | 0 | 0 | 0 | 1
  Discontinued study drug due to adverse event | 3 | 2 | 0 | 3
  Discontinued due to AE related to study drug | 1 | 1 | 0 | 1

25. Secondary Outcome: Percentage of Participants With a Psoriatic Arthritis Response Criteria (PsARC) Response at Week 24
Description: A PsARC response is defined as improvement from Baseline in at least 2 of the following 4 measures, at least 1 of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • At least 30% improvement in the 78 tender joint count, • At least 30% improvement in the 76 swollen joint count, • At least 20% improvement in the patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • At least 20% improvement in the physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Participants with missing data were considered non-responders.
Time Frame: Baseline and Week 24
Population: Participants enrolled in the Extension Phase; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants | 26.1 | 20.0 | 55.0 | 40.0

26. Secondary Outcome: Percentage of Participants With a Modified ACR 20 Response at Week 24
Description: A modified ACR 20 response was defined as a participant who met the following 3 criteria for improvement: • ≥ 20% improvement in 78 tender joint count (includes 10 additional joints often involved in psoriatic arthritis: the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers); • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm VAS); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. Response at Week 24 was measured as improvement from Baseline (Day 1) and from Week 12 (Day 85). Participants with no post-baseline ACR scores were considered non-responders.
Time Frame: Baseline (Day 1), Week 12 (Day 85) and Week 24
Population: Participants enrolled in the Extension Phase; LOCF imputation was used. For the analysis of response from Week 12 (Day 85), participants with a tender or swollen joint count of 0 at Day 85 were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants
  Response From Baseline | 43.5 | 42.5 | 45.0 | 40.0
  Response From Week 12: number analyzed (Participants) | 30 | 34 | 13 | 18
  Response From Week 12 | 16.7 | 14.7 | 15.4 | 16.7

27. Secondary Outcome: Percentage of Participants With a Modified ACR 50 Response at Week 24
Description: A modified ACR 50 response was defined as a participant who met the following 3 criteria for improvement: • ≥ 50% improvement in 78 tender joint count (includes 10 additional joints often involved in psoriatic arthritis: the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers); • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm VAS); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. Response at Week 24 was measured as improvement from Baseline (Day 1) and from Week 12 (Day 85). Participants with no post-baseline ACR scores were considered non-responders.
Time Frame: Baseline (Day 1), Week 12 (Day 85) and Week 24
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants
  Response From Baseline | 23.9 | 22.5 | 20.0 | 15.0
  Response From Week 12: number analyzed (Participants) | 31 | 34 | 13 | 18
  Response From Week 12 | 9.7 | 5.9 | 15.4 | 5.6

28. Secondary Outcome: Percentage of Participants With a Modified ACR 70 Response at Week 24
Description: A modified ACR 70 response was defined as a participant who met the following 3 criteria for improvement: • ≥ 70% improvement in 78 tender joint count (includes 10 additional joints often involved in psoriatic arthritis: the first carpometacarpal [CMC] and the distal interphalangeal [DIP] joints of the fingers); • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm VAS); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. Response at Week 24 was measured as improvement from Baseline (Day 1). Participants with no post-baseline ACR scores were considered non-responders.
Time Frame: Baseline (Day 1) and Week 24
Population: Participants enrolled in the Extension Phase; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants | 13.0 | 17.5 | 15.0 | 5.0

29. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response Based on DAS28-CRP(4) at Week 24
Description: The DAS28 measures the severity of disease at a specific time. DAS28-CRP(4) is derived from the following 4 variables: • 28 tender joint count, (does not include the DIP joints, the hip joint, or the joints below the knee) • 28 swollen joint count • C-reactive protein • Patient's global assessment of disease activity according to the formula: DAS28-CRP(4) = 0.56*√(TJC28) + 0.28*(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96. DAS28 scores range from 0 to 9.4, where higher scores indicate more disease activity. A EULAR response reflects an improvement in disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 > 1.2 from Baseline and attainment of a DAS28 score ≤ 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 > 0.6 and ≤ 1.2 and a DAS28 score ≤ to 5.1 or, • an improvement (decrease) in the DAS28 > 1.2 and a DAS28 score > 3.2
Time Frame: Baseline and Week 24
Population: Participants enrolled in the Extension Phase; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants | 67.4 | 60.0 | 70.0 | 50.0

30. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response Based on DAS28-CRP(3) at Week 24
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: Participants enrolled in the Extension Phase; LOCF imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants | 60.9 | 67.5 | 65.0 | 55.0

31. Secondary Outcome: Maximal ACR Response During the Extension Period
Description: The ACR-N index score was calculated for each participant at each time point in the study according to the following definition: ACR-N = the lowest of the following 3 values: • percent improvement from Baseline in the 76 swollen joint count, • percent improvement from Baseline in the 78 tender joint count • median percent improvement from Baseline in the following 5 measures ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-reactive protein. The maximal ACR-N for each participant during the 12-week extension period was calculated, and represents the maximal ACR response achieved.
Time Frame: ACR was measured at Baseline and Weeks 16, 20 and 24
Population: Participants enrolled in the Extension Phase with non-missing ACR data
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 44 | 39 | 20 | 17
percent improvement | 29.1 (40.86) | 30.4 (36.77) | 23.3 (32.11) | 34.2 (31.16)

32. Secondary Outcome: Time to ACR 20 Response During the Study
Description: Time to ACR 20 was measured from the first dose of apremilast to the first time a participant achieved an ACR 20 response in the treatment or extension phase. The Kaplan-Meier estimates of time to ACR 20 response were calculated for participants who had an ACR 20 response at any time during the study.
Time Frame: Baseline to Week 24
Population: Participants enrolled in the Extension Phase with an ACR 20 response at any time during the study
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 31 | 29 | 4 | 6
days | 43.0 [29.0 to 44.0] | 43.0 [29.0 to 59.0] | 34.0 [29.0 to 55.0] | 55.5 [29.0 to 57.0]

33. Secondary Outcome: Time to ACR 50 Response During the Treatment and Extension Phase
Description: Time to ACR 50 response was measured from the first dose of apremilast to the first time a participant achieved an ACR 50 response in the treatment or extension phase. The Kaplan-Meier estimates of time to ACR 50 response were calculated for participants who had an ACR 50 response at any time during the study.
Time Frame: Baseline to Week 24
Population: Participants enrolled in the Extension Phase with an ACR 50 response at any time during the study
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 18 | 16 | 2 | 3
days | 71.0 [44.0 to 110.0] | 58.5 [56.0 to 86.0] | 84.5 [84.0 to 85.0] | 55.0 [23.0 to 57.0]

34. Secondary Outcome: Time to ACR 70 Response During the Treatment and Extension Phase
Description: Time to ACR 70 response was measured from the first dose of apremilast to the first time a participant achieved an ACR 70 response in the treatment or extension phase. The Kaplan-Meier estimates of time to ACR 70 response were calculated for participants who had an ACR 70 response at any time during the study.
Time Frame: Baseline to Week 24
Population: Participants enrolled in the Extension Phase with an ACR 70 response at any time during the study
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 9 | 7 | 0 | 0
days | 138.0 [85.0 to 169.0] | 85.0 [57.0 to 141.0] |  |

35. Secondary Outcome: Change From Baseline and Week 12 in Dactylitis Severity Score at Week 24
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated on a scale from 0 (no dactylitis) to 3 (severe dactylitis). The dactylitis severity score is the sum of the individual scores for each digit and ranges from 0 to 60. Change in the dactylitis severity score was assessed from Baseline (Day 1) and from Week 12 (Day 85).
Time Frame: Baseline, Week 12 and Week 24
Population: Participants enrolled in the Extension Phase with a baseline/Week 12 value and at least 1 post-baseline value in the extension period; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 39 | 20 | 18
units on a scale
  Change from Baseline | -0.4 (3.47) | -1.5 (3.13) | -1.8 (4.94) | 0.1 (1.08)
  Change from Week 12: number analyzed (Participants) | 45 | 39 | 20 | 18
  Change from Week 12 | 0.3 (3.07) | -0.2 (1.97) | -0.3 (0.98) | -0.8 (2.39)

36. Secondary Outcome: Percentage of Participants With Enthesitis in the Extension Phase
Description: as for outcome 17
Time Frame: Week 12 and Week 24
Population: Participants enrolled in the Extension Phase
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 20
percentage of participants
  Achilles tendon into the calcaneous: Week 12 | 17.4 | 15.0 | 20.0 | 20.0
  Achilles tendon into the calcaneous: Week 24 | 19.6 | 15.0 | 0.0 | 15.0
  Plantar fascia into the calcaneous:Week 12 | 15.2 | 17.5 | 25.0 | 10.0
  Plantar fascia into the calcaneous: Week 24 | 13.0 | 7.5 | 0.0 | 10.0

37. Secondary Outcome: Time to Relapse of Psoriatic Arthritis After Extension Phase
Description: Relapse of psoriatic arthritis was defined as a 50% loss of the maximal ACR improvement during the Follow-up Phase in participants who achieved at least an ACR 20 at their Final Extension Phase (Week 24)/Early Termination Visit. The time to relapse during the Follow-up Phase was calculated from the time of maximum ACR reduction and from the date of the Final Extension Phase visit. Participants classified as responders who did not relapse were censored at the day of the last follow-up.
Time Frame: From Week 24 to the end of the 28-day follow-up (1) and from the date of maximal ACR until the end of the 28-day follow-up phase (2).
Population: Participants with an ACR 20 response at the Week 24 (or Early Termination) visit and entered the Follow-up Phase after the Extension Phase
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 20 | 17 | 2 | 3
days
  1. From Week 12 | 31.0 [29.0 to NA] — Could not be estimated due to the low number of events | 32.0 [29.0 to 38.0] | 16.0 [NA to NA] — Could not be estimated due to the low number of events | 29.0 [15.0 to NA] — Could not be estimated due to the low number of events
  2. From Date of Maximal ACR Response | 85.0 [57.0 to NA] — Could not be estimated due to the low number of events | 111 [41.0 to NA] — Could not be estimated due to the low number of events | 16.0 [NA to NA] — Could not be estimated due to the low number of events | 29.0 [15.0 to NA] — Could not be estimated due to the low number of events

38. Secondary Outcome: Number of Participants Who Relapsed After the Extension Phase
Description: Relapse of psoriatic arthritis was defined as a 50% loss of the maximal ACR improvement during the Follow-up Phase in participants who achieved at least an ACR 20 at their Final Extension Phase/Early Termination Visit.
Time Frame: Week 24 to Week 28 (28-day follow-up period)
Population: as for outcome 37
Measure: Number; unit: participants
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 20 | 17 | 2 | 3
participants | 8 | 8 | 1 | 2

39. Secondary Outcome: Change From Baseline and Week 12 in SF-36 at Week 24
Description: as for outcome 20
Time Frame: Baseline (Day 1), Week 12 (Day 85) and Week 24
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 43 | 36 | 20 | 18
units on a scale
  Mental Component: Change from Baseline: number analyzed (Participants) | 41 | 36 | 20 | 18
  Mental Component: Change from Baseline | 0.2 (9.08) | 1.4 (8.92) | -2.7 (12.20) | -1.0 (14.00)
  Mental Component: Change from Week 12: number analyzed (Participants) | 43 | 34 | 20 | 18
  Mental Component: Change from Week 12 | -1.1 (8.14) | -2.4 (9.35) | -2.5 (10.60) | -3.4 (10.61)
  Physical Component: Change from Baseline: number analyzed (Participants) | 41 | 36 | 20 | 18
  Physical Component: Change from Baseline | 3.2 (6.68) | 4.4 (7.74) | 1.8 (9.50) | 4.2 (9.99)
  Physical Component: Change from Week 12: number analyzed (Participants) | 43 | 34 | 20 | 18
  Physical Component: Change from Week 12 | 0.3 (6.10) | 1.0 (6.60) | -0.1 (8.50) | 2.5 (7.81)

40. Secondary Outcome: Change From Baseline and Week 12 in Dermatology Life Quality Index (DLQI) at Week 24
Description: The DLQI is a validated, self-administered, 10-item questionnaire that measures the impact of skin disease on participants' quality of life, based on recall over the past week. Domains include symptoms, feelings, daily activities, leisure, work, personal relationships, and treatment. Each question is answered on a scale from 0 (not at all) to 3 (very much) The total score ranges from 0 to 30 where a higher score indicates that a participant's dermatological condition has a greater impact on their daily life.
Time Frame: Baseline (Day 1), Week 12 (Day 85) and Week 24
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 43 | 37 | 20 | 18
units on a scale
  Change from Baseline | -3.0 (7.36) | -1.5 (4.08) | -2.6 (4.78) | -1.9 (5.50)
  Change from Week 12 | -0.0 (5.72) | -0.1 (3.54) | -1.2 (2.07) | -2.0 (6.25)

41. Secondary Outcome: Change From Baseline and Week 12 in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 24
Description: as for outcome 22
Time Frame: Baseline (Day 1), Week 12 (Day 85) and Week 24
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 46 | 40 | 20 | 18
units on a scale
  Change from Baseline | -0.1 (0.45) | -0.2 (0.37) | -0.1 (0.61) | -0.2 (0.59)
  Change from Week 12: number analyzed (Participants) | 46 | 40 | 20 | 17
  Change from Week 12 | 0.0 (0.37) | -0.0 (0.23) | -0.0 (0.46) | -0.2 (0.44)

42. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy for Fatigue (FACIT-F) at Week 24
Description: as for outcome 23
Time Frame: Baseline (Day 1), Week 12 (Day 85) and Week 24
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 40 mg QD | Apremilast 20 mg BID | Placebo/Apremilast 40 mg QD | Placebo/Apremilast 20 mg BID
Number analyzed (Participants) | 43 | 37 | 20 | 18
units on a scale
  Change from Baseline | 4.4 (9.76) | 5.9 (7.76) | 1.3 (11.23) | 1.3 (12.34)
  Change from Week 12 | -0.3 (8.56) | 0.1 (6.19) | -2.4 (9.05) | -1.3 (13.10)

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the 12-week placebo-controlled phase, including AEs that occurred during the 28-day observational follow-up, and for up to 24 weeks for all participants who were randomized or re-randomized to apremilast at any time during the study.
Groups:
- Week 12: Apremilast 40 mg QD: Participants received 40 mg apremilast once daily (QD) for 12 weeks during the Treatment Phase.
- Week 12: Apremilast 20 mg BID: Participants received 20 mg apremilast twice a day (BID) for 12 weeks during the Treatment Phase.
- Week 12: Placebo: Participants received matching placebo to apremilast for 12 weeks during the Treatment Phase.
- Week 24: Apremilast 40 mg QD: Participants who received 40 mg QD apremilast, regardless of when the apremilast exposure started (at Week 0, or 12), up until Week 24.
- Week 24: Apremilast 20 mg BID: Participants who received 20 mg apremilast BID, regardless of when the apremilast exposure started (at Week 0, 12), up until Week 24.
Arm/Group | Week 12: Apremilast 40 mg QD | Week 12: Apremilast 20 mg BID | Week 12: Placebo | Week 24: Apremilast 40 mg QD | Week 24: Apremilast 20 mg BID
Serious Adverse Events (participants affected / at risk) | 0/67 | 4/69 | 6/68 | 3/87 | 8/89
Other Adverse Events (participants affected / at risk) | 45/67 | 44/69 | 42/68 | 63/87 | 62/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Week 12: Apremilast 40 mg QD (N=67) | Week 12: Apremilast 20 mg BID (N=69) | Week 12: Placebo (N=68) | Week 24: Apremilast 40 mg QD (N=87) | Week 24: Apremilast 20 mg BID (N=89)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 1 | 0 | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Week 12: Apremilast 40 mg QD (N=67) | Week 12: Apremilast 20 mg BID (N=69) | Week 12: Placebo (N=68) | Week 24: Apremilast 40 mg QD (N=87) | Week 24: Apremilast 20 mg BID (N=89)
Nasopharyngitis (Infections and infestations) | 8 | 8 | 14 | 23 | 18
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 0 | 4 | 3
Influenza (Infections and infestations) | 3 | 0 | 1 | 5 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0 | 5
Headache (Nervous system disorders) | 15 | 13 | 11 | 17 | 17
Dizziness (Nervous system disorders) | 7 | 3 | 3 | 7 | 3
Migraine (Nervous system disorders) | 2 | 6 | 0 | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 18 | 14 | 7 | 23 | 14
Nausea (Gastrointestinal disorders) | 15 | 12 | 10 | 23 | 14
Abdominal pain upper (Gastrointestinal disorders) | 4 | 7 | 3 | 5 | 8
Vomiting (Gastrointestinal disorders) | 4 | 4 | 3 | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 1 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 1 | 5 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 4 | 6
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 5 | 7 | 8 | 10 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 4 | 1
Fatigue (General disorders) | 11 | 6 | 6 | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.